CLINICAL TRIAL: NCT05348694
Title: OsteoPreP: The Effect of Probiotic Supplementation on Bone, Muscle, and Glucose Metabolism in Postmenopausal Women: A Randomised Placebo-controlled Trial
Brief Title: OsteoPreP: Food Supplements for Postmenopausal Bone Health
Acronym: OsteoPreP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Australian Catholic University (Other)
Collaborators: Pendulum Therapeutics (Industry); Curtin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-122HC
Record Dates: First submitted 2022-04-18; First posted 2022-04-27 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-01

CONDITIONS: Postmenopausal Osteopenia; Bone Loss, Age Related; Age-Related Sarcopenia; Glucose Metabolism Disorders; Age-related Cognitive Decline
Keywords: Postmenopausal bone loss; Probiotics; Volumetric bone mineral density; Short-chain fatty acids
MeSH Terms: conditions — Osteoporosis; Glucose Metabolism Disorders; Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pendulum WBF-038 (Active Comparator): Pendulum WBF-038, a proprietary formulation of the following strains: Akkermansia muciniphila, Clostridium butyricum, Clostridium beijerinckii, Anaerobutyricum hallii, Bifidobacterium infantis, plus chicory inulin and magnesium stearate - 1 capsule with the morning meal and 1 capsule with the evening meal for 12 months.
  Interventions: Dietary Supplement: Pendulum WBF-038
- Pendulum Placebo (Placebo Comparator): Pendulum Placebo containing Magnesium stearate - 1 capsule with the morning meal and 1 capsule with the evening meal for 12 months.
  Interventions: Dietary Supplement: Pendulum Placebo

INTERVENTIONS:
Dietary Supplement: Pendulum WBF-038 — All bacteria contained in Pendulum WBF-038 are commensal organisms that have been repeatedly documented to inhabit the human gastrointestinal tract under normal circumstances. Pendulum's WBF-038 is a proprietary formulation of the following strains: Akkermansia muciniphila, Clostridium butyricum, Clostridium beijerinckii, Anaerobutyricum hallii, Bifidobacterium infantis, plus chicory inulin and magnesium stearate. The organisms were grown under controlled conditions consistent with Good Manufacturing Practices (GMP) and employ no animal-derived products. All ingredients utilized during manufacturing were food grade and qualified as generally recognized as safe (GRAS).
  The product is provided as acid-resistant capsules in bottles that are to be stored refrigerated at 4℃.
  Arms: Pendulum WBF-038
Dietary Supplement: Pendulum Placebo — Pendulum placebo capsules containing magnesium stearate
  Arms: Pendulum Placebo

SUMMARY:
To evaluate the effect of 12 months of supplementation with a probiotic (probiotic plus prebiotic; 2 capsules per day) on relative change (%) in total volumetric bone density (measured using high resolution peripheral quantitative computed tomography [HR-pQCT]) of the distal tibia.

DETAILED DESCRIPTION:
It is well established that bone loss occurs throughout life after the attainment of peak bone mass which is usually reached by the end of the second decade of life. During the first 5-8 years following menopause, women experience an accelerated bone loss, which is then followed by a slower phase of decline in bone mineral density (BMD). As over 40% of all women in Australia will suffer an osteoporotic (fragility) fracture in their lifetime, investigating interventions that can prevent bone loss in postmenopausal women is a critical focus. The menopausal transition is also associated with an increased risk of cardiovascular disease, diabetes, and cognitive decline. These conditions and their treatments can also affect bone health.

Previous research has indicated a potential link between the gut microbiome and bone health. Animal studies indicate that interventions affecting the gut microbiome may be successful in reducing bone loss, but human data is limited. Moreover, there is an emerging body of evidence linking the gut microbiome to cognitive, muscle and cardiometabolic function. Such studies indicate that probiotics (healthy gut bacteria) or prebiotics (food for healthy bacteria, e.g. fibre) can increase the amount of short chain fatty acids - such as butyrate -produced by the bacteria in the gut which may mediate the beneficial effects of improving gut health.

The proposed study is a double-blind, placebo-controlled randomised trial, which will investigate whether consuming a probiotic supplement containing inulin (a prebiotic soluble fibre) twice daily for 12 months will improve bone health in postmenopausal women. In addition, secondary outcomes will measure the effect of the intervention on immune system modulation and cognition as well as musculoskeletal and metabolic function as potential mediators.

One hundred and sixty postmenopausal women residing in Melbourne (Victoria, Australia) who are at least one year from their final menses will be recruited from the community via a mail out, advertisements in newspapers, social media, flyers as well as a landing page on an ACU managed website. The investigators have also applied for assisted mail outs through Services Australia for recruitment purposes. Services Australia is able to extract names and addresses of some target study demographics (females living in Melbourne aged between 40 and 65) from the Medicare database and mail them the study details on our behalf. Those wishing to participate will undergo a series of baseline assessments inclusive of bone mineral density scans, blood and stool sampling and physical activity and lifestyle questionnaires. They will then be randomised, in a blinded fashion, to consume one of the following two supplements:

* Placebo control group (n = 80): Placebo capsule - 2 capsules per day
* Probiotics group (n=80): Probiotic capsule - 2 capsules per day

Study outcomes will be measured at baseline, 6 months, and 12 months. In addition, participants will be contacted via the telephone and email at three-month and nine-month timepoints to report any adverse responses to the supplementation. At the 12-month time point, participants will cease supplementation and immediately (within 24 hours) attend a post intervention assessment and will complete identical assessment measures to those they did at baseline. Finally, at 2 weeks post supplementation cessation participants will be asked to attend an appointment to provide a final stool sample.

If it can be confirmed that long term consumption of a probiotic supplement can have beneficial effects on bone health, muscle health, and metabolic health in postmenopausal women, this intervention could be recommended in the prevention of osteoporosis and associated musculoskeletal and metabolic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, 40-65 years old
* Caucasian (due to significant differences in BMD and bone remodelling between ethnicities)
* At least one year since final menses
* Signed informed consent
* Up to date Covid 19 vaccination status
* Able to walk without the use of an aid
* Stated availability throughout the entire study period
* Mental capacity to understand and willingness to fulfil all the details of the protocol
* Residing in Melbourne, Victoria, Australia

Exclusion Criteria:

* Diagnosis of osteoporosis
* T-score of -2.5 or less at the femoral neck or lumbar spine (L1-L4) on the DXA scan at screening visit
* HbA1c ≥6.5% at screening visit
* Blood pressure at screening visit of systolic >180 mmHg and/or diastolic >120 mmHg
* Untreated hyperthyroidism
* Rheumatoid arthritis
* Diagnosed with a disease-causing secondary osteoporosis or malabsorption: chronic obstructive pulmonary disease, inflammatory bowel disease, celiac disease, type 1/type 2 diabetes, or chronic liver disease
* Bariatric surgery
* Recently diagnosed malignancy (within the last 5 years)
* Current or recent oral corticosteroid use (any dose within the last 3 months, or 5mg of Prednisolone (or equivalent) or a higher daily dose for 14 days or more 3-12 months prior to screening)
* Use of antiresorptive therapy, including systemic hormone replacement therapy, bisphosphonates, strontium ranelate (current or during the last 3 years)
* Use of teriparatide (current or during the last 3 years)
* Participation in other clinical intervention trials
* Antibiotics treatment 2 months prior to inclusion
* Unwilling to cease taking other probiotic or prebiotic supplements (current use)

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — OsteoPreP is an intervention trial for the prevention of bone loss in early post-menopausal women
Enrollment: 160 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Total volumetric bone mineral density of the distal tibia | 12 months
  Percentage change in total volumetric bone density measured using high resolution peripheral quantitative computed tomography (HR-pQCT) of the distal tibia.

SECONDARY OUTCOMES:
Bone mineral density of the lumbar spine | 12 months
  Relative change in lumbar spine (L1-L4) bone mineral density (BMD) measured using dual energy X-ray absorptiometry (DXA)
Bone mineral density of the hip | 12 months
  Relative change in total hip BMD measured using DXA
Tibia and radius trabecular bone volume | 12 months
  Relative change in tibia and radius trabecular bone volume fraction measured using HR-pQCT
Tibia and radius cortical area | 12 months
  Relative change in tibia and radius cortical area measured using HR-pQCT
Tibia and radius cortical volumetric bone mineral density | 12 months
  Relative change in tibia and radius cortical volumetric BMD measured using HR-pQCT
Total volumetric bone mineral density of the distal radius | 12 months
  Relative change in total volumetric BMD of the distal radius measured using HRpQCT
Serum C-terminal cross-linking telopeptide of type I collagen (ßCTX-I) - bone turnover marker | 6 months and 12 months
  Relative change in ßCTX-I in serum
Serum procollagen type 1 N-terminal propeptide (P1NP) - bone turnover marker | 6 months and 12 months
  Relative change in P1NP levels in serum
Serum osteocalcin (OC) - bone turnover marker | 6 months and 12 months
  Relative change in OC in serum
Short-chain fatty acids (SCFAs) | 6 months, 12 months, and 2 weeks post intervention
  Relative change in SCFA levels (including butyrate) in stool
16s rRNA genetic sequencing of the gut microbiota | 6 months, 12 months, and 2 weeks post intervention
  Relative change in species-level gut microbiota composition in stool using 16s rRNA sequencing
Fasting blood glucose | 6 months and 12 months
  Relative change in fasted blood glucose levels in circulating blood
Glycated haemoglobin (HbA1c) | 6 months and 12 months
  Relative change in HbA1c levels in circulating blood
Lower leg muscle area | 12 months
  Relative change in lower leg muscle area measured using HR-pQCT
Lean body mass | 12 months
  Relative change in appendicular lean body mass measured using DXA
Grip strength | 6 months and 12 months
  Relative change in left and right hand grip strength measured using a hand dynamometer
High-sensitivity C-reactive protein (hs-CRP) | 6 months and 12 months
  Relative change in hs-CRP levels in serum
Regulatory T lymphocytes (Tregs) | 12 months
  Relative change in circulating number of Tregs in blood
Oral glucose tolerance test (OGTT) | 6 months and 12 months
  Relative change in oral glucose tolerance in circulating blood
Muscle tissue glycogen content | 6 months and 12 months
  Relative change in muscle tissue glycogen content obtained from a muscle biopsy
Muscle tissue triglyceride content | 6 months and 12 months
  Relative change in muscle tissue triglyceride content obtained from a muscle biopsy
Muscle tissue type 1 fibre composition | 6 months and 12 months
  Relative change in muscle tissue type 1 fibre proportion obtained from a muscle biopsy
Lipocalin2 | 6 months, 12 months, and 2 weeks post intervention
  Relative change in Lipocalin2 (intestinal inflammation) in stool
Cogstate One back Test Cognitive performance test | 6 months and 12 months
  Relative change in speed of performance and number of errors in the One Back Test using the Cogstate cognitive assessment tool. Lower score = better performance
Cogstate Groton Maze Learning Test Cognitive performance test | 6 months and 12 months
  Relative change in number of errors in the Groton Maze Learning Test using the Cogstate cognitive assessment tool. Lower score = better performance
Cogstate Continuous Paired Associate Learning Test Cognitive performance test | 6 months and 12 months
  Relative change in accuracy of performance and number of errors in the Continuous Paired Associate Learning Test using the Cogstate cognitive assessment tool. Lower score = better performance
Cogstate Social Emotional Cognition Test Cognitive performance test | 6 months and 12 months
  Relative change in accuracy of performance in the Social Emotional Cognition Test using the Cogstate cognitive assessment tool. Higher score = better performance
Depression, Anxiety and Stress Scale 21 | 6 months and 12 months
  Relative change in depression, anxiety and stress measured using the Depression Anxiety and Stress Scale 21 (DASS-21) questionnaire. The DASS-21 has a minimum score of 0 and a maximum score of 63 with higher scores indicating a worse outcome.
Gastrointestinal Symptom Rating Scale | 6 months and 12 months
  Relative change in gastrointestinal symptoms measured using the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire. The GSRS has a minimum score of 5 and a maximum score of 45 with higher scores indicating a worse outcome.
Plasma glucagon-like peptide 1 | 6 months and 12 months
  Relative change in gut hormone glucagon-like peptide 1 [GLP-1] in plasma
Plasma peptide tyrosine-tyrosine | 6 months and 12 months
  Relative change in gut hormone peptide tyrosine-tyrosine [PYY] in plasma
Plasma adiponectin | 6 months and 12 months
  Relative change adiponectin in plasma
EuroQol Five Dimensions Quality of life Medical Outcome Survey | 6 months and 12 months
  Relative change in quality of life measured using the EuroQol Five Dimensions (EQ-5D) questionnaire. The EQ-5D has a minimum score of Level 1 and a maximum score of Level 5 with higher levels indicating a worse outcome
Social Interaction Anxiety Scale | 6 months and 12 months
  Relative change in social anxiety measured using the Social Interaction Anxiety Scale (SIAS) questionnaire. The SIAS has a minimum score of 0 and a maximum score of 80 with higher scores indicating a worse outcome.
The Warwick-Edinburgh Mental Wellbeing Scale | 6 months and 12 months
  Relative change in mental wellbeing measured using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) questionnaire. The WEMWBS has a minimum score of 14 and a maximum score of 70 with higher scores indicating a better outcome.
Continuous blood glucose level monitoring for 10 days | 6 months and 12 months
  Relative change in blood glucose (area under the curve) over 10 days measured using a continuous glucose monitoring device
Fasting blood insulin | 6 months and 12 months
  Relative change in fasted blood insulin levels in circulating blood
Fat mass | 12 months
  Relative change in total body fat mass measured using DXA
Blood metabolomics | 12 months
  Relative change in blood metabolites using liquid chromatography-mass spectrometry
Office blood pressure | 6 months and 12 months
  Relative change in Systolic and Diastolic blood pressure measured using a sphygmomanometer
The Visual Analogue Scale Pain Intensity | 6 months and 12 months
  Relative change in current pain intensity measured using a visual analogue scale (VAS) pain intensity scale. The VAS has a minimum score of 0 and a maximum score of 10 with higher scores indicating a worse outcome.
Calprotectin | 6 months, 12 months, and 2 weeks post intervention
  Relative change in calprotectin (intestinal inflammation) in stool
Muscle mass | 12 months
  Relative change in total body muscle mass measured using DXA

CONTACTS AND LOCATIONS:
Overall Officials: John Hawley, PhD, Principal Investigator — Australian Catholic University
Locations (1):
- Australian Catholic University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turbic A, Vandenput L, Gandham A, Lorentzon M. Effects of Synbiotic Supplementation on Bone and Metabolic Health in Caucasian Postmenopausal Women: Rationale and Design of the OsteoPreP Trial. Nutrients. 2024 Dec 6;16(23):4219. doi: 10.3390/nu16234219. PMID 39683612